CLINICAL TRIAL: NCT05405205
Title: Effect of a Synbiotic on Body Fat Mass, Weight Management, Traits of Metabolic Syndrome and Gut Permeability in Individuals With Abdominal Overweight: a Randomised, Controlled, Double-blind Clinical Study
Brief Title: Effect of Synbiotic L. Fermentum Strains on Body Fat Mass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Slimbiotics GmbH (Industry)
Collaborators: Clinical Research Center Kiel GmbH (Other)
Responsible Party: Sponsor
Organization: Slimbiotics (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Slim-LfX2-2021
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Weight, Body
Keywords: synbiotic; probiotic; body fat mass; abdominal overweight
MeSH Terms: conditions — Body Weight | interventions — Synbiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All three products are identical in smell, flavour, color, texture, appearance, packaging (sachets) and labelling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- synbiotic (Experimental): synbiotic consisting of three different strains of Lactobacillus fermentum + acacia gum (gum arabic)
  Interventions: Dietary Supplement: synbiotic
- probiotic (Experimental): probiotic consisting of the identical three different strains of Lactobacillus fermentum
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: synbiotic — Consumption of 6 g powder consisting of the strains Lactobacillus fermentum K7-Lb1, L. fermentum K8- Lb1, L. fermentum K11-Lb3, acacia gum (gum arabic), maltodextrin, sucralose and flavour twice a day resolved in drinking water
  Arms: synbiotic
Dietary Supplement: probiotic — Consumption of 6 g powder consisting of the strains Lactobacillus fermentum K7-Lb1, L. fermentum K8- Lb1, L. fermentum K11-Lb3, maltodextrin, sucralose and flavour twice a day resolved in drinking water
  Arms: probiotic
Dietary Supplement: placebo — Consumption of 6 g powder containing microcrystalline cellulose, maltodextrin , sucralose and flavour twice a day, resolved in drinking water
  Arms: placebo

SUMMARY:
In this placebo-controlled trial the effect of a synbiotic consisting of three different strains of Lactobacillus fermentum and acacia gum (gum arabic) was compared with a probiotic formulation containing identical strains on body fat mass, body weight management, traits of metabolic syndrome and gut permeability in individuals who are abdominally overweight.

DETAILED DESCRIPTION:
The effects of probiotics on glucose and lipid metabolism, on body fat, weight, visceral fat and liver steatosis were shown by several meta-analyses for the total variety, as described above. Some probiotic species/strains, however, seem to be more efficacious (Koutnikova et al., 2019). The lactobacilli used in this trial were selected for their anti-inflammatory properties and based on induction of defensins in enterocytes. Therefore, one may expect more pronounced effects of these strains on traits of the metabolic syndrome, which is driven by low grade inflammation, than those found in the meta-analyses for the whole variety of probiotics without discriminating species and strain specificity.

The combination of these Lactobacillus strains with acacia gum is expected to enable even more pronounce effects, since acacia gum was shown to increase the number of lactobacilli in the gut (Cherbut et al., 2003; Calame et al., 2008) and, hence, are supposed to promote their propagation and, hence their effects. The dosage of 10 g/day acacia gum was demonstrated to be sufficient for enhancing fecal lactobacilli and bifidobacterial (Cherbut et al., 2003; Calame et al., 2008).

Acacia gum, however, seems to have own effects on traits of the metabolic syndrome. Even though the effects still need to be confirmed in more DB-RCTs, one may suggest a separate effect, e.g. by reduction of the SGLT1in the intestine (Nasir et al., 2010).

This DB-RCT aims at providing first evidence for an effect of this symbiotic on traits of the metabolic syndrome. The target parameters were selected for allowing a health claim according to the Health Claim Directive of the EU (REGULATION (EC) No 1924/2006 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 20 December 2006 on Nutrition and Health Claims Made on Foods) and/or the REGULATION (EU) No 609/2013 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 12 June 2013 for Food for Special Medical Purposes after having confirmative evidence.

The following health claim options are feasible according to the EFSA Guidance on the scientific requirements for health claims related to appetite ratings, weight management, and blood glucose concentrations (EFSA Journal 2012;10(3):2604) and to the EFSA Guidance on the scientific requirements for health claims related to antioxidants, oxidative damage and cardiovascular health (EFSA Journal 2011;9(12):2474):

* Beneficial effect on long-term glycemia (glucose metabolism) as assessed by HbA1c,
* facilitates weight management as assessed by body weight, BMI, waist circumference, or body fat mass,
* reduces insulin resistance, a risk factor for type 2 diabetes, as assessed by HOMA-IR,
* reduces LDL-C, a risk factor coronary heart disease,
* increases HDL-C, a beneficial physiological effect. It is noteworthy that EFSA admits demonstration of effects in type 2 diabetes for health claims on these target parameters assuming that there is a continuity of these parameters from healthy to impaired metabolism (EFSA Journal 2012;10(3):2604).

Alternatively, the following claims may be used as FSMPs:

* For dietary management of impaired glucose metabolism and type 2 diabetes
* for dietary weight management in overweight
* for dietary management of insulin resistance The primary parameter has been selected by estimating the sample size for these potential targets based on the most recent meta-analysis of Koutnikova et al. 2019. Since we expect a more pronounced effect by the selected strains and the combination with acacia gum (see above) we assumed a twofold higher effect than found for the whole variety of probiotics. Taking this into account, the target parameter with the lowest estimated sample size was body fat in individuals with type 2 diabetes (N = 56 for each arm). Accordingly, this target was defined as primary parameter.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI ≥ 25)
* Elevated waist circumference (>94cm and >80cm (for European men and women, respectively)
* Age ≥ 18
* Written informed consent

Exclusion Criteria:

* Subjects currently enrolled in another clinical study
* Subjects having finished another clinical study within the last 4 weeks before inclusion
* Hypersensitivity, allergy or intolerance against any compound of the test products (e. g. acacia gum)
* Condition after implantation of a cardiac pacemaker or other active implants
* Sulfonylurea treatment
* Any disease or condition which might compromise significantly the hepatic (ascites), hematopoietic, renal, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system with the exception of the conditions defined by the inclusion criteria
* History of or present liver deficiency as defined by Quick < 70%
* Regular medical treatment including OTC, which may have impact on the study aims (e. g. probiotics containing supplements, laxatives, steroids etc.)
* History of hepatitis B, C, HIV
* Major cognitive or psychiatric disorders
* Subjects who are scheduled to undergo any diagnostic intervention or hospitalization which may cause protocol deviations
* Simultaneous study participation by members of the same household
* Pregnancy and lactation
* Ascites as assessed by sonography
* Any diet to lose body weight
* Eating disorders or vegan diet
* Anorexic drugs
* Present drug abuse or alcoholism
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Body Fat Mass | 12 weeks
  Body Fat Mass (BFM) as assessed by bioelectrical impedance analysis (BIA) (alteration V3-V1; synbiotic versus placebo

SECONDARY OUTCOMES:
Visceral Adiposity Index | 12 weeks
  Visceral Adiposity Index (VAI) after Amato et al. Diabetes Care 33:920-922, 2010: (Females: VAI = WC / (36.58 + (1.89 × BMI)) × (TG/0.81) × (1.52/HDL)), (Males: VAI = (WC / (39.68 + (1.88 × BMI)) × (TG/1.03) × (1.31/HDL)

OTHER OUTCOMES:
HOMA-IR | 12 weeks
  HOMA-IR (Homeostasis Model Assessment (HOMA)-IR = glucose [mmol/L] x insulin [μU/ml]/22,5) as parameter for insulin resistance
MSX-index | 12 weeks
  MSX-index (alteration V3-V1) according to ATP III/IDF* definitions (Waist x FPG x Tg x 1/HDL-C x BPsys x BPdias) (ascites as interfering cause for alteration of these measures will be excluded by abdominal sonography)
Sagittal abdominal diameter (SAD) | 12 weeks
  Sagittal abdominal diameter (SAD): Distance between the under surface of the rectus muscle and the anterior wall of the aorta - measure for visceral fat after Armellini et al. 1991: Sagittal abdominal diameter as a practical predictor of visceral fat, Int J Obes. 1991

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Essl, Study Director — Slimbiotics GmbH
Locations (1):
- Clincal Research Center Kiel GmbH, Kiel, Schleswig-Holstein, Germany